CLINICAL TRIAL: NCT04012762
Title: The Acute Responses of Muscles Properties to the Different Whole Body Vibration Training
Brief Title: Vibration Training and Muscles Properties
Acronym: CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tülay Çevik (Other)
Responsible Party: Sponsor-Investigator, Tülay Çevik, Principal Investigator, Okan University
Organization: Okan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Bitlis Eren University
Record Dates: First submitted 2019-07-08; First posted 2019-07-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Muscle Relaxation
Keywords: Muscle Power, Muscle Flexibility, Muscle Tone, Whole-Body Vibration Training.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderate-intensity group (Active Comparator): WBVT application was 2-4 mm for vibration amplitude value and 25 Hz for training frequency in moderate-intensity group.
  Interventions: Device: Whole body vibration training
- Vigorous-intensity group (Active Comparator): WBVT application was 2-4 mm for vibration amplitude value and 40 Hz for training frequency in vigorous-intensity group.
  Interventions: Device: Whole body vibration training

INTERVENTIONS:
Device: Whole body vibration training — Intermittent whole-body vibration exposure is a training method providing physical stimulation effect on skeletal muscles by increasing gravitational acceleration on the vibration platform.

SUMMARY:
Application dose standards have not yet been determined for Whole Body Vibration Training which is subject to studies with different frequencies and amplitudes. Our objective was to examine acute responses of two different vibration training doses on muscle tone, strength, and flexibility.

DETAILED DESCRIPTION:
Application dose standards have not yet been determined for Whole Body Vibration Training which is subject to studies with different frequencies and amplitudes. Our objective was to examine acute responses of two different vibration training doses on muscle tone, strength, and flexibility.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and untrained participants.
* Dominant side of the participants was recorded and only right dominant individuals were included.

Exclusion Criteria:

* Participants with body weight over 120 kg.
* Participants had lower extremity trauma and lower extremity movement restriction.
* Participants who had any cardiovascular or neurological conditions, dizziness or vertigo

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Muscle Tone | 30 minute
  Tone assessments were made by MyotonPro Digital Palpation Device.
Muscle power | 30 minute
  The muscle power evaluation was made by Lafayette Manuel Muscle Testing System.
Flexibility | 30 minute
  Hamstring flexibility was evaluated with Sit and Reach Test.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Atıcı, Ph. D., Principal Investigator — Okan University
Locations (1):
- Okan University, Tuzla, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No